CLINICAL TRIAL: NCT00595686
Title: A Phase 1, Open-label, Dose-Escalation Study Of The Safety And Pharmacokinetics Of SNX-5422 Mesylate In Subjects With Refractory Hematological Malignancies
Brief Title: Safety And Pharmacology Of SNX-5422 Mesylate In Subjects With Refractory Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esanex Inc. (Industry)
Collaborators: Serenex, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1311002; SNX-5422-CLN1-002
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Hematologic Neoplasms
Keywords: Hematologic Malignancies Hsp90 Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — SNX-5422

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: SNX-5422

INTERVENTIONS:
Drug: SNX-5422 — dose escalated; tablets every other day; undetermined duration until disease progression

SUMMARY:
Hsp90 is a chemical in the body that is involved in the promotion of cancer. SNX-5422 is an experimental drug that blocks Hsp90. It is being evaluated for safety and efficacy in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Karnofsky performance status > 60
* confirmed hematological malignancy
* refractory to available therapy or for which no therapy is available
* adequate hepatic, renal and hematological function

Exclusion Criteria:

* CNS malignancy
* at risk for prolonged QT interval
* significant GI/liver disease
* other serious concurrent illness or medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
adverse events and other safety assessments | continuous

SECONDARY OUTCOMES:
disease response specific to the hematological malignancy | after every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Nashville, Tennessee

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1311002&StudyName=Safety%20And%20Pharmacology%20Of%20SNX-5422%20Mesylate%20In%20Subjects%20With%20Refractory%20Hematological%20Malignancies